CLINICAL TRIAL: NCT04051957
Title: Isosorbide Mononitrate For Anti-Vascular Endothelial Growth Factor (VEGF) Induced Kidney Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Delays due to COVID and loss of research coordinator.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, Jaya Kala, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-19-0429
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Results first posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Kidney Injury; Proteinuria; Hypertension
Keywords: Kidney Injury; Proteinuria; Hypertension; Anti-VEGF
MeSH Terms: conditions — Proteinuria; Hypertension | interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isosorbide Mononitrate (Experimental)
  Interventions: Drug: Isosorbide Mononitrate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Isosorbide Mononitrate — The starting dose will be Isosorbide Mononitrate 60 mg ER daily and after 4 weeks, if tolerated but response is not achieved, the dose will be escalated to Isosorbide Mononitrate 120 mg ER daily (2 tabs of 60 mg ER tablets).
  Arms: Isosorbide Mononitrate
Drug: Placebo oral tablet — Placebo will be given daily and will be doubled after 4 weeks of start of therapy.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the hypothesis that isosorbide mononitrate prevents deterioration of renal function in patients receiving anti-angiogenic therapies that target vascular endothelial growth factor (VEGF).

ELIGIBILITY:
Inclusion Criteria:

* Patients on or enrolled for anti-VEGF therapy
* new-onset proteinuria, defined as a urine protein: creatinine ratio (UPC) of >500mg/g or hypertension (Systolic BP ≥ 140 mm Hg and/or diastolic BP ≥ 90 mm Hg) or a decrease in eGFR by ≥ 25% from baseline before starting therapy.

Exclusion Criteria:

* Pregnant women
* Breast-feeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaya Kala, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University Of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Isosorbide Mononitrate | Placebo
Started | 7 | 2
Completed | 5 | 2
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isosorbide Mononitrate | Placebo | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 2 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 6 | 2 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction in Urine Protein Creatinine Ratio (UPC) of > 500 mg/Day From That Measured Before Enrollment
Time Frame: Baseline, Month 1
Population: Data were not collected for 2 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 5 | 2
Participants | 1 | 0

2. Primary Outcome: Number of Participants With a Reduction in UPC of > 500 mg/Day From That Measured Before Enrollment
Time Frame: Baseline, Month 2
Population: Data were not collected for 2 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 5 | 2
Participants | 1 | 0

3. Primary Outcome: Number of Participants With a Reduction in UPC of > 500 mg/Day From That Measured Before Enrollment
Time Frame: Baseline, Month 3
Population: Data were not collected for 2 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 5 | 2
Participants | 3 | 1

4. Secondary Outcome: Number of Participants With Improvement in Estimated Glomerular Filtration Rate (eGFR) ≥25% From Before Enrollment
Time Frame: Baseline, Month 1
Population: Data were not collected for 2 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 5 | 2
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Improvement in Estimated Glomerular Filtration Rate (eGFR) ≥25% From Before Enrollment
Time Frame: Baseline, Month 2
Population: Data were not collected for 2 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 5 | 2
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Improvement in Estimated Glomerular Filtration Rate (eGFR) ≥25% From Before Enrollment
Time Frame: Baseline, Month 3
Population: Data were not collected for 2 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 5 | 2
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 1
Population: Data were not collected for 3 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 4 | 2
Participants | 0 | 1

8. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 2
Population: Data were not collected for 3 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 4 | 2
Participants | 2 | 1

9. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 3
Population: Data were not collected for 3 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 4 | 2
Participants | 3 | 1

10. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 4
Population: Data were not collected for 2 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 5 | 2
Participants | 4 | 2

11. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 5
Population: Data were not collected for 3 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 4 | 2
Participants | 2 | 1

12. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 6
Population: Data were not collected for 3 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 4 | 2
Participants | 3 | 2

13. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 7
Population: Data were not collected for 3 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 4 | 2
Participants | 3 | 2

14. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 8
Population: Data were not collected for 2 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 5 | 2
Participants | 3 | 2

15. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 9
Population: Data were not collected for 3 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 4 | 2
Participants | 3 | 2

16. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 10
Population: Data were not collected for 3 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 4 | 2
Participants | 2 | 2

17. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 11
Population: Data were not collected for 3 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 4 | 2
Participants | 3 | 2

18. Secondary Outcome: Number of Participants With Reduction in Systolic Blood Pressure (SBP) of ≥ 10 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 5 mm Hg From Before Enrollment
Time Frame: Baseline, Week 12
Population: Data were not collected for 2 in the Isosorbide Mononitrate arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate | Placebo
Number analyzed (Participants) | 5 | 2
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Isosorbide Mononitrate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 2/7 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isosorbide Mononitrate (N=7) | Placebo (N=2)
Dizziness (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to the COVID pandemic and limited clinical face-to-face appointments leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT04051957/Prot_001.pdf